CLINICAL TRIAL: NCT02907853
Title: Combating Craving With Contingency Management: Neuroplasticity and Methamphetamine Abuse in South Africa
Brief Title: Contingency Management for Meth in South Africa Methamphetamine Abuse in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21CMinSA; NCT02948868 (obsolete NCT alias)
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contingency Management (Experimental): In exchange for consecutive urine samples documenting methamphetamine abstinence, participants receive increasingly valuable reinforcers.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — as described above

SUMMARY:
This study will link findings from neuroscience with clinical outcomes using contingency management (CM) to identify changes in brain structure and function that emerge during purely behavioral therapy for methamphetamine (MA) use.

DETAILED DESCRIPTION:
This study will correlate MA-abstinence outcomes from an 8-week program of voucher-based incentives using an escalating schedule for 30 treatment-seeking, MA-dependent individuals with scores on tasks of working memory and assessments of neuropsychological and demographic status. At the beginning and end of the CM program, participants will participate in MRI scans while performing a working memory task and will complete a battery of select neurocognitive and psychological assays to address two specific aims: (1) to determine whether changes in neural function within frontostriatal circuitry from baseline to end of the 8-week CM program are associated with parallel changes in measures of cognitive control and impulsivity and with MA abstinence outcomes and (2) to determine whether structural changes in frontostriatal circuitry over the 8-week CM intervention correspond with neurocognitive, psychological and MA abstinence measures.

ELIGIBILITY:
Inclusion Criteria:

* provide voluntary informed consent
* meet DSM-5 criteria for MA or amphetamine use disorder
* provide at least one urine sample positive for MA/amphetamine metabolites during screening (i.e. prior to the commencement of the study).
* aged 18-45
* right-handed
* English-speaking

Exclusion Criteria:

* currently receiving treatment for stimulant addiction or needing more intensive treatment than outpatient care
* meet DSM-5 criteria for substance use disorder other than nicotine
* unable to attend 4+ visits during the 2-week screening period or to complete measures
* Physical or mental illness that would require intervention that would alter imaging or that would interfere with safe study participation
* pregnant, claustrophobic, or have metal prostheses, cardiac pacemakers, or metal clips that are incompatible with the scanner
* HIV positive status
* unable to comprehend written or spoken English
* currently taking psychiatric medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Responses to Contingency Management | 8 weeks
  urine samples documenting methamphetamine abstinence
fMRI Measures | Change b/w baseline and 8 Weeks
  measures of resting state connectivity

SECONDARY OUTCOMES:
Stop Signal Task | Change b/w baseline and 8 Weeks
  measure of inhibitory control
Continuous Performance Task | Change b/w baseline and 8 Weeks
  test of sustained attention
Stroop | Change b/w baseline and 8 Weeks
  test of inhibitory control
Balloon Analog Risk Task | Change b/w baseline and 8 Weeks
  measure of risk taking and decision making

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry at Groote Schuur Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other investigators following publication of the main paper or 2 years after the last subject completes participation, whichever comes first. Shared data will be stripped of all PHI and potentially personally identifying variables.
  Requests should briefly state the concept of interest, provide a brief timeline for analyzing the data and preparing a manuscript, and include a copy of the CV of the investigator making the request and documentation of proof of training in the ethical treatment of human subjects in research.
  The concept proposal will be evaluated based on three criteria, including the potential impact or contribution to the research in advancing knowledge; the feasibility of the proposed research; and that the aim of the proposed research will not overlap with any of the aims or planned analyses.